CLINICAL TRIAL: NCT04841343
Title: Randomized Controlled Trial of Triamcinolone Impregnated Hemostatic Bioabsorbable Middle Meatus Nasal Packing Following Endoscopic Sinus Surgery
Brief Title: Triamcinolone Packing Following Endoscopic Sinus Surgery
Status: Completed | Type: Observational
Sponsor: University of California, Los Angeles (Other)
Responsible Party: Principal Investigator, Marilene Wang, Principal Investigator, University of California, Los Angeles
Other Study IDs: 20-002080
Record Dates: First submitted 2021-04-07; First posted 2021-04-12 (Actual); Last update posted 2023-08-01 (Actual); Status verified 2023-07

CONDITIONS: Sinusitis
MeSH Terms: conditions — Sinusitis | interventions — Triamcinolone

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

INTERVENTIONS:
Drug: Triamcinolone — Triamcinolone in sinus

SUMMARY:
Endoscopic sinus surgery (ESS) is a well-established treatment strategy for medically refractory chronic rhinosinusitis. Middle meatus spacers are currently used following ESS to prevent scarring, synechiae formation, and middle turbinate lateralization. A 2012 systematic review favored spacers compared to no spacers, with a follow up 2013 systematic review finding no difference between the use of absorbable and non-absorbable spacers. This review, however, noted that steroidal spacers may reduce middle meatus scarring and adhesions. More recent data has shown the effectiveness of steroid releasing middle meatus implants in preventing middle turbinate lateralization, reducing synechiae formation, and reducing revision surgery. However, these stents are costly, and may result in excess crusting postoperatively, which limits their use in some settings. Another study investigated the use of steroid-impregnated absorbable packing materials, and demonstrated the safety and utility of this method of middle meatus packing. However, a limitation to this study was overall low enrollment with only 19 total patients enrolled.

The purpose of this project is to add to the existing body of evidence regarding middle meatus spacers, by studying the impact of steroid impregnated, bioabsorbable hemostatic packing (Hemopore®, Stryker) on postoperative visualization and scar formation.

DETAILED DESCRIPTION:
Introduction

Endoscopic sinus surgery (ESS) is a well-established treatment strategy for medically refractory chronic rhinosinusitis. Middle meatus spacers are currently used following ESS to prevent scarring, synechiae formation, and middle turbinate lateralization. A 2012 systematic review favored spacers compared to no spacers, with a follow up 2013 systematic review finding no difference between the use of absorbable and non-absorbable spacers. This review, however, noted that steroidal spacers may reduce middle meatus scarring and adhesions. More recent data has shown the effectiveness of steroid releasing middle meatus implants in preventing middle turbinate lateralization, reducing synechiae formation, and reducing revision surgery. However, these stents are costly, and may result in excess crusting postoperatively, which limits their use in some settings. Another study investigated the use of steroid-impregnated absorbable packing materials, and demonstrated the safety and utility of this method of middle meatus packing. However, a limitation to this study was overall low enrollment with only 19 total patients enrolled.

The purpose of this project is to add to the existing body of evidence regarding middle meatus spacers, by studying the impact of steroid impregnated, bioabsorbable hemostatic packing (Hemopore®, Stryker) on postoperative visualization and scar formation.

Research Design The proposed study will be a randomized controlled trial comparing steroid impregnated bioabsorbable and dissolvable nasal packing to non-steroid impregnated packing. Potential subjects will be adults, aged 18 and older, with a diagnosis of chronic rhinosinusitis based on the 2016 International Consensus Statement on Allergy and Rhinology: Rhinosinusitis definition, who have failed a trial of previous medical therapy, have bilateral sinus disease on CT imaging, and will undergo bilateral endoscopic sinus surgery. If the patient chooses to proceed with surgery for their medically refractory chronic rhinosinusitis they will be introduced to the research proposal and if willing to participate, the informed consent process will take place, during their preoperative visit. On the day of surgery the patient's right and left sinuses will be randomized to either steroid or no steroid middle meatus packing. At the end of the surgical procedure, the attending surgeon will soak the Hemopore in either 5 cc Duobiotic saline irrigation (bacitracin 50,000 units, polymyxin B 500,000 units in 0.9% sodium chloride 500mL) or 1 ml of triamcinolone 40 mg/ml (Kenalog-40, Bristol-Myers Squibb) mixed with 5 cc Duobiotic saline irrigation and label them 1 (no steroid) and 2 (steroid). The fellow or resident surgeon will then insert the packing into the middle meatus, with the steroid packing going into the side randomized for steroid, and the non-steroid packing going into the other side. A password protected data file will be maintained in UCLA Box, accessible to the investigators, where the side of placement of the packing will be recorded. Postoperative visits will be scheduled at the usual time points: 7-10 days, 24-30 days, and 2-3 months post-op. Nasal endoscopy will be performed at each visit, as a standard post op procedure. Video recording of the endoscopy will be saved for review at the conclusion of the study for determination of the patency of the postop cavity using the Lund-Kennedy endoscopic scoring system (LKES) and the perioperative sinus endoscopy (POSE) score . Symptom scores will also be collected and reviewed, as it is current practice for patients to respond to the sinonasal outcome test-22 (SNOT-22) at preop and postop visits. LKES and POSE scores will be recorded in a password protected file in UCLA Box that is separate from the file containing the side of steroid packing.

The investigators plan to enroll 50 consecutive patients in this study, over the course of about 4-6 months. At the end of the study period, the endoscopy scores (LKES and POSE) will be compared between the steroid and non-steroid sides. Each patient will serve as his/her own control. Statistical analysis will be performed using paired t tests for continuous variables and chi-square tests for categorical variables. A p value < 0.05 will be considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* aged 18 and older
* diagnosis of chronic rhinosinusitis based on the 2016 International Consensus Statement on Allergy and Rhinology: Rhinosinusitis definition
* failed a trial of previous medical therapy
* have bilateral sinus disease on CT imaging
* will undergo bilateral endoscopic sinus surgery.

Exclusion Criteria:

* unable to give informed consent
* not a candidate for endoscopic sinus surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients over age 18 who have bilateral chronic sinusitis who have failed previous medical therapy and will undergo endoscopic sinus surgery
Sampling Method: Non-Probability Sample
Enrollment: 22 (Actual)
Dates: Start 2021-01-29 (Actual); Primary Completion 2021-09-30 (Actual); Study Completion 2022-09-30 (Actual)

PRIMARY OUTCOMES:
Lund Kennedy Endoscopy score | 1 week
  Assessment of inflammation, crusting, polyps, edema in sinus; Scale from 0 to 2, with higher scores meaning worse outcome

CONTACTS AND LOCATIONS:
Locations (1):
- UCLA Medical Center, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Zhao X, Grewal A, Briel M, Lee JM. A systematic review of nonabsorbable, absorbable, and steroid-impregnated spacers following endoscopic sinus surgery. Int Forum Allergy Rhinol. 2013 Nov;3(11):896-904. doi: 10.1002/alr.21201. Epub 2013 Jul 24. PMID 23894058
- [Result] Cote DW, Wright ED. Triamcinolone-impregnated nasal dressing following endoscopic sinus surgery: a randomized, double-blind, placebo-controlled study. Laryngoscope. 2010 Jun;120(6):1269-73. doi: 10.1002/lary.20905. PMID 20513050